CLINICAL TRIAL: NCT03840798
Title: Disseminating Child Abuse Clinical Decision Support to Improve Detection, Evaluation and Reporting
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); University of Wisconsin, Madison (Other); Northwell Health (Other)
Responsible Party: Principal Investigator, Rachel Berger MD, MPH, Professor of Pediatrics and Clinical and Translational Science, Chief, Division of Child Advocacy, University of Pittsburgh
Other Study IDs: PRO18010135; DI-2017C1-6215 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2019-01-07; First posted 2019-02-15 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Child Abuse; Physical Abuse; Trauma; Child Maltreatment
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pretest/Baseline period
- Posttest/go-live period
  Interventions: Other: Child Abuse Clinical Decision Support system

INTERVENTIONS:
Other: Child Abuse Clinical Decision Support system — The investigators are implementing the following aspects of the Electronic Health Record (EHR) based child abuse- clinical decision support (CA-CDS) system.
  1. a universal child abuse screen (CAS)
  2. an embedded child abuse alert system
  3. alerts to physicians and advanced practice providers
  4. physical abuse order sets
  Groups: Posttest/go-live period

SUMMARY:
Child maltreatment is a leading cause of death and disability in children. More than 3 million reports to Child Protective Services are made every year in the US and almost 1,600 children die annually due to maltreatment. Children who are victims of maltreatment often have significant lifelong adverse health, social, and economic consequences.

Accurate and timely recognition of the early signs of child maltreatment is critical to decreasing morbidity and mortality. A significant proportion of children who suffer severe morbidity and/or mortality from maltreatment had been previously evaluated by physician(s) who did not recognize the abuse. The American Academy of Pediatrics has evidence-based recommendations for the testing which should be done as part of the medical evaluation of children with suspected physical abuse. However, despite these evidence-based recommendations, physicians fail to consistently screen for and evaluate for abuse even in high-risk situations.

The investigators have developed and evaluated what the investigators believe to be the first, comprehensive electronic health record (EHR) based child abuse clinical decision support (CA-CDS). This EHR-based CA-CDS system informs medical care at multiple points during the care for a potentially maltreated child, beginning with identification of suspected abuse to the handing off of information to CPS which has a mandate to protect children who are victims of suspected maltreatment.

The investigators are disseminating the following aspects of the Electronic Health Record (EHR) based child abuse- clinical decision support (CA-CDS) system which they developed as part of the investigator's initial PCORI grant.

1. a universal child abuse screen (CAS) - supports identification of maltreatment
2. an embedded child abuse alert system - supports identification of maltreatment
3. alerts to physicians and advanced practice providers - supports identification of maltreatment
4. physical abuse order set - supports proper evaluation of suspected physical abuse
5. documentation assistance for making reports of suspected maltreatment to Child Protective Services - supports mandated reporting

The primary objective is to disseminate and implement CA-CDS in two different EHRs in two hospital systems - Northwell Health (NY) and University of Wisconsin (WI) - and to assess whether the CA-CDS improves identification, evaluation and mandated reporting of child maltreatment.

Aim #1 is to compare the rates of identification of possible child abuse - defined as reports to Child Protective Services - before and after integration of CA-CDS into the EHR among children presenting to 5 Emergency Departments in two different health systems.

Aim #2 is to compare the rate of physician compliance with American Academy of Pediatrics guidelines for evaluation of suspected physical abuse before and after integration of CA-CDS into the EHR in 5 Emergency Departments in two health care systems.

Once the D&I is complete, the investigators will have demonstrated the feasibility of implementing the CA-CDS in the three EHRs which make up 85% of all the US EHRs. This is a critical step towards the goal of having a CA-CDS as a standard EHR component.

DETAILED DESCRIPTION:
Child maltreatment is a leading cause of death and disability in children. More than 3 million reports to Child Protective Services are made every year in the US and almost 1,600 children die annually due to maltreatment. Children who are victims of maltreatment often have significant lifelong adverse health, social, and economic consequences.

Accurate and timely recognition of the early signs of child maltreatment is critical to decreasing morbidity and mortality. A significant proportion of children who suffer severe morbidity and/or mortality from maltreatment had been previously evaluated by physician(s) who did not recognize the abuse. The American Academy of Pediatrics has evidence-based recommendations for the testing which should be done as part of the medical evaluation of children with suspected physical abuse. However, despite these evidence-based recommendations, physicians fail to consistently screen for and evaluate for abuse even in high-risk situations.

The investigators have developed and evaluated what the investigators believe to be the first, comprehensive electronic health record (EHR) based child abuse clinical decision support (CA-CDS). This EHR-based CA-CDS system informs medical care at multiple points during the care for a potentially maltreated child, beginning with identification of suspected abuse to the handing off of information to CPS which has a mandate to protect children who are victims of suspected maltreatment.

The investigators are disseminating the following aspects of the Electronic Health Record (EHR) based child abuse- clinical decision support (CA-CDS) system which they developed as part of the investigator's initial PCORI grant.

1. a universal child abuse screen (CAS) - supports identification of maltreatment
2. an embedded child abuse alert system - supports identification of maltreatment
3. alerts to physicians and advanced practice providers - supports identification of maltreatment
4. physical abuse order set - supports proper evaluation of suspected physical abuse
5. documentation assistance for making reports of suspected maltreatment to Child Protective Services - supports mandated reporting

The primary objective is to disseminate and implement CA-CDS in two different EHRs in two hospital systems - Northwell Health (NY) and University of Wisconsin (WI) - and to assess whether the CA-CDS improves identification, evaluation and mandated reporting of child maltreatment.

Aim #1 is to compare the rates of identification of possible child abuse - defined as reports to Child Protective Services - before and after integration of CA-CDS into the EHR among children presenting to 5 Emergency Departments in two different health systems.

Aim #2 is to compare the rate of physician compliance with American Academy of Pediatrics guidelines for evaluation of suspected physical abuse before and after integration of CA-CDS into the EHR in 5 Emergency Departments in two health care systems.

Process metrics: Rapid cycle usability testing will be one of the earliest assessments of the end-user acceptability of the CA-CDS and changes will be made to the CA-CDS based on these data. Process metrics which will be measured throughout the live period, including proportion of patients who receive a CAS, how often the CAS is positive, which question(s) of the CAS are positive, how often any part of the CA-CDS triggers, how often order sets are used, and how often providers dismiss the alert.

Short-term outcomes: Descriptive statistics will be used to describe the demographics of the population. For Aim 1, the primary outcome is the report made to CPS. The proportion of children who have a report made to CPS will be calculated for both the silent mode (before) and live (after) groups, including race and insurance type. For Aim 2, the primary outcome is compliance with the AAP guidelines for evaluation of suspected abuse in children <2 yrs of age. The proportion of providers who are compliant with the guidelines will be calculated for both groups. Another short-term outcome will be the use of provider surveys to determine the impact of the CA-CDS on clinical decision making and efficacy with identifying and evaluating suspected child maltreatment. The investigators will also evaluate the impact of provider training and patient racial, ethnic and socioeconomic status on these outcomes.

Long-term outcomes: A long-term outcome is whether the CA-CDS is integrated into clinical practice after the end of the D&I. Another long-term outcome is evaluation of the proportion of cases of child maltreatment in which the child had been evaluated at least once previously and the diagnosis of abuse was missed; a decrease in this proportion is a true measure of improved outcome.

Once the D&I is complete, the investigators will have demonstrated the feasibility of implementing the CA-CDS in the three EHRs which make up 85% of all the US EHRs. This is a critical step towards the goal of having a CA-CDS as a standard EHR component.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to one of the partner hospitals AND age less than 10 years old at Wisconsin site OR age less than 13 at Northwell site

Exclusion Criteria:

* None

Max Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children who present to one of the participating emergency departments during the baseline or go-live periods
Sampling Method: Non-Probability Sample
Enrollment: 351 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Change in the number of reports made to Child Protective Services (CPS) | Up to 52 weeks for the baseline period, up to 52 weeks for the go-live period
  Number of reports to CPS made in baseline compared to go-live periods
Change in the compliance with American Academy of Pediatrics guidelines for evaluation of suspected abuse in patients <2 years of age | Up to 52 weeks for the baseline period, up to 52 weeks for the go-live period
  Percent compliance with American Academy of Pediatrics guidelines for evaluation of suspected abuse in patients <2 years of age during the baseline period compared to go-live period

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Berger, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Northwell Health, Manhasset, New York
  - University of Wisconsin, Madison, Wisconsin